CLINICAL TRIAL: NCT01736137
Title: Evaluation of the Six Minute Walk Test, Heart Rate Variability and Quality of Life in Heart Failure Patients on Beta-blocker Treatment
Brief Title: Evaluation of the Six Minute Walk Test and Other Instruments in Heart Failure
Status: Completed | Type: Observational
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Débora Lara Zuza Scheucher, Physiotherapist, Federal University of Uberlandia
Other Study IDs: dont have
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Heart Failure; Autonomic Nervous System Imbalance; Heart Rate and Rhythm Disorders; Quality of Life
Keywords: Heart failure; Autonomic Nervous System; Heart rate; Quality of life
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic Heart failure group: All chronic heart failure group participants will perform two walk tests at the same day, with a heart rate monitor, and answer questionnaires about their perception of quality of life. Tests will be conducted on a single day, without follow up of patients. The six minute walk test will be performed according the American Thoracic Society Statement (2002).
  Interventions: Other: Six minute walk test
- Control Group: All control group participants will perform two walk tests at the same day, with a heart rate monitor, and answer questionnaires about their perception of quality of life. Tests will be conducted on a single day, without follow up of patients. The six minute walk test will be performed according the American Thoracic Society Statement (2002).
  Interventions: Other: Six minute walk test

INTERVENTIONS:
Other: Six minute walk test — If patients meet the criteria of the study, their data will be collected and will be interviewed to fill the Minnesota Living with Heart Failure Questionnaire (MLHFQ). They then will be taken to the hallway to perform the six minute walk test monitored with a heart rate monitor (Polar RS800 CX). After the test there will be a break of 20 to 30 minutes before repeating the walk test. During rest time, the patient will answer the general health survey questionnaire: Medical Outcome Study 36-item Short-Form Health Survey (SF-36).
  Other Names: MLHFQ; SF-36; Heart rate variability (Polar RS800 CX)

SUMMARY:
The purpose of this study is to assess functional capacity, quality of life and functioning of the autonomic nervous system in heart failure patients on beta-blocker treatment. The study hypothesis is that subjects who walk less distance, have lower quality of life and reduced heart rate variability during the six minute walk test.

DETAILED DESCRIPTION:
Heart failure and its treatment result in symptoms such as pulmonary or systemic congestion causing impairment to the effort, psychological and social commitment, and impact on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Different etiologies of Heart Failure
* Functional class I - III (NYHA)
* Left ventricular ejection fraction (LVEF) ≤ 50%
* No history of previous cardiac surgery
* In return for medical evaluation at the Amelio Marques Clinic, Hospital de Clinicas, Federal University of Uberlândia scheduled for the period from October 2012 to January 2013
* Clinical stability observed by: heart rate, respiratory rate, blood pressure and arterial oxygen saturation

Exclusion Criteria:

* Bad cognition compromising the understanding of tests
* Physical disability that compromise the performance in walk test
* Aortic aneurysm or any aortic deformity
* Patients with signs or symptoms of transient myocardial ischemia with angina pectoris and/or class IV by the Canadian Cardiovascular Society Classification
* Anomalous pressure behavior with hypertension > 180/100 mmHg
* Orthostatic hypotension (decrease > 15 mmHg ) with symptoms
* Arrhythmia with presence of complex ventricular extra systoles
* Tachycardia sinus at rest (HR > 120 beats/min)
* Atrioventricular block of 2nd or 3rd degree
* Subjects with pacemakers or implantable cardioverter-defibrillator (ICD)
* Functional class IV by the New York Heart Association
* Chronic organ dysfunction such as renal failure, respiratory or liver disease
* Active neoplasia over the past five years
* Commitment as general weakness, fever, other limiting factors (psychological, musculoskeletal)
* Feeling sick before the beginning of the Six minute walk test: intolerable angina or dyspnea, cramps in legs, staggering gait, excessive sweating (diaphoresis), pallor or ashen skin or SpO2 below 85%
* Voluntary desire of the patient to withdraw from research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Heart failure patients routinely treated at the Amelio Marques Clinic, Hospital de Clínicas, Federal University of Uberlandia, who have scheduled a visit during the period of study and attends the criterias of the study will be included.
  The sample will be a convenience, and included all patients who meet the study criteria.
  The control group included healthy participants with the same gender and age of the chronic heart failure group.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2011-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Maximum distance walked | During six minute walk test
  The six minute walk test will be performed twice by each patient, at the same day. The collection period will extend until the sample is complete. This is an observational study because there is no follow up and reassessment of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Celia R Lopes, PhD, Study Chair — Federal University of Uberlandia
Locations (1):
- Amelio Marques Clinic, Uberlândia, Minas Gerais, Brazil

REFERENCES:
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Bocchi EA, Braga FG, Ferreira SM, Rohde LE, Oliveira WA, Almeida DR, Moreira Mda C, Bestetti RB, Bordignon S, Azevedo C, Tinoco EM, Rocha RM, Issa VS, Ferraz A, Cruz Fd, Guimaraes GV, Montera Vdos S, Albuquerque DC, Bacal F, Souza GE, Rossi Neto JM, Clausell NO, Martins SM, Siciliano A, Souza Neto JD, Moreira LF, Teixeira RA, Moura LZ, Beck-da-Silva L, Rassi S, Azeka E, Horowitz E, Ramires F, Simoes MV, Castro RB, Salemi VM, Villacorta Junior H, Vila JH, Simoes R, Albanesi F, Montera MW; Sociedasde Brasileira de Cardiologia. [III Brazilian Guidelines on Chronic Heart Failure]. Arq Bras Cardiol. 2009;93(1 Suppl 1):3-70. No abstract available. Portuguese. PMID 20963312
- [Background] Bocchi EA, Marcondes-Braga FG, Bacal F, Ferraz AS, Albuquerque D, Rodrigues Dde A, Mesquita ET, Vilas-Boas F, Cruz F, Ramires F, Villacorta H Jr, Souza Neto JD, Rossi Neto JM, Moura LZ, Beck-da-Silva L, Moreira LF, Rohde LE, Montera MW, Simoes MV, Moreira Mda C, Clausell N, Bestetti R, Mourilhe-Rocha R, Mangini S, Rassi S, Ayub-Ferreira SM, Martins SM, Bordignon S, Issa VS. [Updating of the Brazilian guideline for chronic heart failure - 2012]. Arq Bras Cardiol. 2012 Jan;98(1 Suppl 1):1-33. doi: 10.1590/s0066-782x2012001000001. No abstract available. Portuguese. PMID 22392082
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Reis MS, Deus AP, Simoes RP, Aniceto IA, Catai AM, Borghi-Silva A. Autonomic control of heart rate in patients with chronic cardiorespiratory disease and in healthy participants at rest and during a respiratory sinus arrhythmia maneuver. Rev Bras Fisioter. 2010 Mar-Apr;14(2):106-13. Epub 2010 May 7. English, Portuguese. PMID 20464168
- [Background] Carvalho VO, Guimaraes GV, Carrara D, Bacal F, Bocchi EA. Validation of the Portuguese version of the Minnesota Living with Heart Failure Questionnaire. Arq Bras Cardiol. 2009 Jul;93(1):39-44. doi: 10.1590/s0066-782x2009000700008. English, Portuguese, Spanish. PMID 19838469
- [Background] Dantas RA, Sawada NO, Malerbo MB. [Research on quality of life: review of the scientific production of public universities from the state of Sao Paulo]. Rev Lat Am Enfermagem. 2003 Jul-Aug;11(4):532-8. doi: 10.1590/s0104-11692003000400017. Portuguese. PMID 14748173
- [Background] Enright PL, McBurnie MA, Bittner V, Tracy RP, McNamara R, Arnold A, Newman AB; Cardiovascular Health Study. The 6-min walk test: a quick measure of functional status in elderly adults. Chest. 2003 Feb;123(2):387-98. doi: 10.1378/chest.123.2.387. PMID 12576356
- [Background] Faggiano P, D'Aloia A, Gualeni A, Brentana L, Dei Cas L. The 6 minute walking test in chronic heart failure: indications, interpretation and limitations from a review of the literature. Eur J Heart Fail. 2004 Oct;6(6):687-91. doi: 10.1016/j.ejheart.2003.11.024. No abstract available. PMID 15542403
- [Background] [I National Consensus of Cardiovascular Rehabilitation]. Arq Bras Cardiol. 1997 Oct;69(4):267-91. No abstract available. Portuguese. PMID 9595722
- [Background] Guazzi M, Dickstein K, Vicenzi M, Arena R. Six-minute walk test and cardiopulmonary exercise testing in patients with chronic heart failure: a comparative analysis on clinical and prognostic insights. Circ Heart Fail. 2009 Nov;2(6):549-55. doi: 10.1161/CIRCHEARTFAILURE.109.881326. Epub 2009 Sep 28. PMID 19919979
- [Background] Guyatt GH, Sullivan MJ, Thompson PJ, Fallen EL, Pugsley SO, Taylor DW, Berman LB. The 6-minute walk: a new measure of exercise capacity in patients with chronic heart failure. Can Med Assoc J. 1985 Apr 15;132(8):919-23. PMID 3978515
- [Background] Moura LZ, Guimaraes GV, Pires PV, Cruz F, Stopa G, Bocchi EA. Exercise chemosensitivity in heart failure: ventilatory, chronotropic and neurohormonal responses. Arq Bras Cardiol. 2010 Sep;95(3):381-91. doi: 10.1590/s0066-782x2010005000110. Epub 2010 Aug 13. PMID 20721516
- [Background] Opasich C, Pinna GD, Mazza A, Febo O, Riccardi R, Riccardi PG, Capomolla S, Forni G, Cobelli F, Tavazzi L. Six-minute walking performance in patients with moderate-to-severe heart failure; is it a useful indicator in clinical practice? Eur Heart J. 2001 Mar;22(6):488-96. doi: 10.1053/euhj.2000.2310. PMID 11237544
- [Background] Pinsky MR. Cardiovascular issues in respiratory care. Chest. 2005 Nov;128(5 Suppl 2):592S-597S. doi: 10.1378/chest.128.5_suppl_2.592S. PMID 16306058
- [Background] Rajendra Acharya U, Paul Joseph K, Kannathal N, Lim CM, Suri JS. Heart rate variability: a review. Med Biol Eng Comput. 2006 Dec;44(12):1031-51. doi: 10.1007/s11517-006-0119-0. Epub 2006 Nov 17. PMID 17111118
- [Background] Santos RD; Sociedade Brasileira de Cardiologia. [III Brazilian Guidelines on Dyslipidemias and Guideline of Atherosclerosis Prevention from Atherosclerosis Department of Sociedade Brasileira de Cardiologia]. Arq Bras Cardiol. 2001 Nov;77 Suppl 3:1-48. No abstract available. Portuguese. PMID 11781591
- [Background] Sparrow J, Parameshwar J, Poole-Wilson PA. Assessment of functional capacity in chronic heart failure: time-limited exercise on a self-powered treadmill. Br Heart J. 1994 Apr;71(4):391-4. doi: 10.1136/hrt.71.4.391. PMID 8198895
- [Result] Bittner V, Weiner DH, Yusuf S, Rogers WJ, McIntyre KM, Bangdiwala SI, Kronenberg MW, Kostis JB, Kohn RM, Guillotte M, et al. Prediction of mortality and morbidity with a 6-minute walk test in patients with left ventricular dysfunction. SOLVD Investigators. JAMA. 1993 Oct 13;270(14):1702-7. PMID 8411500
- [Result] Carvalho EE, Costa DC, Crescencio JC, Santi GL, Papa V, Marques F, Schmidt A, Marin-Neto JA, Simoes MV, Gallo Junior L. Heart failure: comparison between six-minute walk test and cardiopulmonary test. Arq Bras Cardiol. 2011 Jul;97(1):59-64. doi: 10.1590/s0066-782x2011005000056. Epub 2011 May 6. English, Portuguese, Spanish. PMID 21552646
- [Result] Correa FR, da Silva Alves MA, Bianchim MS, Crispim de Aquino A, Guerra RL, Dourado VZ. Heart rate variability during 6-min walk test in adults aged 40 years and older. Int J Sports Med. 2013 Feb;34(2):111-5. doi: 10.1055/s-0032-1321888. Epub 2012 Sep 12. PMID 22972244
- [Result] Enright PL, Sherrill DL. Reference equations for the six-minute walk in healthy adults. Am J Respir Crit Care Med. 1998 Nov;158(5 Pt 1):1384-7. doi: 10.1164/ajrccm.158.5.9710086. PMID 9817683
- [Result] Rector TS, Cohn JN. Assessment of patient outcome with the Minnesota Living with Heart Failure questionnaire: reliability and validity during a randomized, double-blind, placebo-controlled trial of pimobendan. Pimobendan Multicenter Research Group. Am Heart J. 1992 Oct;124(4):1017-25. doi: 10.1016/0002-8703(92)90986-6. PMID 1529875
- [Result] da Silva MA, Sousa AG, Schargodsky H. [Risk factors for acute myocardial infarction in Brazil. FRICAS Study]. Arq Bras Cardiol. 1998 Nov;71(5):667-75. Portuguese. PMID 10347949